CLINICAL TRIAL: NCT07397689
Title: Sepsis Optimal Recognition Toolkit in Children (SORT): An Early Recognition Tool for Children in Asia
Brief Title: Early Sepsis Recognition Tool
Acronym: SORT
Status: Not yet recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Chong Shu-Ling, Dr, KK Women's and Children's Hospital
Other Study IDs: 2023-2640; HCSAINV25jan-0001 (Other Grant/Funding Number: National Medical Research Council)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Infection; Sepsis
Keywords: Phoenix sepsis score; early recognition; infection; child
MeSH Terms: conditions — Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: ARM 1: Retrospective cohort study of children hospitalised with suspected infection from 1st January 2020 to 31st December 2025, among participating sites of the Pediatric Acute & Critical Care Medicine Asian Network (PACCMAN).
  Interventions: Other: Application of the Phoenix Sepsis Score
- Prospective Cohort: ARM 2: Prospective cohort study of children hospitalised with suspected infection from 1st February 2026 to 30th June 2028, among participating sites of the Pediatric Acute & Critical Care Medicine Asian Network (PACCMAN)
  Interventions: Other: Application of the Phoenix Sepsis Score

INTERVENTIONS:
Other: Application of the Phoenix Sepsis Score — Data Variables in the first 24 hours of hospital admission as per Phoenix Sepsis Score: Including that of respiratory function (PaO2:FiO2 and SpO2:FiO2 ratios, need for oxygen, high-flow, non-invasive or mechanical ventilation support), cardiovascular function (including need for vasoactive medications, lactate value and mean arterial pressure), coagulopathy (measured using platelets, International Normalized Ratio, D-dimer and Fibrinogen), neurologic dysfunction (measured with Glasgow Coma Scale and presence of fixed pupils), endocrine (blood glucose), immunologic (absolute neutrophil and absolute lymphocyte count), renal (creatinine levels) and hepatic (total bilirubin and alanine transaminase). Data from the Emergency Departments will need to be linked to inpatient records to obtain the worst values in each domain that occurred in the first 24 hours.

SUMMARY:
This study seeks to develop early recognition tools specially designed for children meeting the Phoenix definition and explore implementation science aspects by investigating facilitators and barriers to adopting Phoenix sepsis criteria in clinical practice. This addresses the critical need for systemic, evidence-based approaches to paediatric sepsis identification across diverse healthcare settings in Asia.

DETAILED DESCRIPTION:
SPECIFIC AIMS AND HYPOTHESES Specific Aim 1: Among children < 18 years old with suspected infection hospitalised in participating Pediatric Acute & Critical Care Medicine Asian Network sites, the investigators seek to compare mortality risk among those with a Phoenix sepsis score of ≥ 2 against those with a score < 2.

Hypothesis 1: The investigators hypothesize that that in-hospital mortality (%) will increase at least 5-times in both higher-resource and lower-resource sites when children with suspected infection have a Phoenix sepsis score of ≥ 2 (compared to those with a score of <2). This is based on published Phoenix data.

Specific Aim 2: The investigators aim to derive and validate the Sepsis Optimal Recognition Toolkit in children (SORT) among children (< 18 years old) with suspected infection in both higher-resource and lower-resource sites in the Pediatric Acute and Critical Care Medicine in Asia Network (PACCMAN).

Hypothesis 2: The investigators hypothesize that SORT will perform with a sensitivity of 90% and a c-statistic of at least 0.80 in predicting for sepsis as defined by a Phoenix Sepsis Score ≥ 2.

Specific Aim 3: The investigators seek to understand the feasibility and acceptability of implementing the Phoenix criteria across PACCMAN sites.

Hypothesis 3: The investigators hypothesize that the parameters required by the Phoenix sepsis score will be feasible and that clinicians and patients will find it acceptable to apply in routine practice.

Exploratory Aim: The investigators aim to study the mimickers of sepsis among children < 18 years old with a Phoenix sepsis score of ≥ 2.

Hypothesis (Exploratory): The investigators hypothesize that children with tissue hypoperfusion from cardiac, hypovolemia and toxicology causes will fulfil Phoenix criteria and mimic sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Children < 18 years old
* Suspected infection defined by (1) blood culture performed (irrespective of result), AND (2) use of broad-spectrum anti-microbial agents, in the first 24 hours of admission

Exclusion Criteria:

* 18 years and older
* Patients who discharge At Own Risk (AOR) without outcome data

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children < 18 years old with suspected infection. Suspected infection is defined as children who undergo blood cultures and receive broad-spectrum anti-microbial agents in the first 24 hours of admission. Anti-microbial agents include antibiotics, antiviral, antifungal and antimalarial medications.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Performance of Phoenix Sepsis Score in Pediatric Acute and Critical Care Medicine in Asia Network (PACCMAN) sites in Asia | 2 years
  Following Specific Aim 1: The primary outcome measure is to validate the Phoenix Sepsis Score in PACCMAN sites in Asia, with the clinical outcome of Mortality. The performance will be measured using area under the receiver operating characteristic curve (AUROC).
Performance of Phoenix Sepsis Score in Pediatric Acute and Critical Care Medicine in Asia Network (PACCMAN) sites in Asia | 2 years
  Following Specific Aim 1: The primary outcome measure is to validate the Phoenix Sepsis Score in PACCMAN sites in Asia, with the clinical outcome of Mortality. The performance will be measured using area under precision recall curve (AUPRC).
  We will also measure the performance using sensitivity, specificity, positive and negative predictive values.
Derivation of an early recognition tool called Sepsis Optimal Recognition Toolkit in children (SORT) | 2 years
  Following the second specific Aim, the outcome is for the model SORT to be derived with a sensitivity of 90% and a c-statistic of at least 0.80 in predicting for sepsis as defined by a Phoenix Sepsis Score ≥ 2.

CONTACTS AND LOCATIONS:
Locations (19):
- Shanghai Children's Medical Center, Shanghai Jiaotong University, Shanghai, China
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong
- Malaysia (8):
  - Hospital Pulau Pinang, George Town
  - Hospital Sultanah Aminah Johor Bahru, Johor Bahru
  - Hospital Tengku Ampuan Rahimah, Klang
  - Hospital Tunku Azizah (Hospital Wanita dan Kanak-Kanak Kuala Lumpur), Kuala Lumpur
  - UKM: Hospital Tunku Ampuan Besar Tuanku Aishah Rohani, Kuala Lumpur
  - University Malaya Medical Centre (UMMC), Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Hospital Sultan Idris Shah, Serdang
- Aga Khan University, Karachi, Pakistan
- King Abdullah Specialist Children's Hospital, Riyadh, Saudi Arabia
- Singapore (2):
  - KK Women's and Children' Hospital, Singapore
  - National University Hospital, Singapore
- Taiwan (2):
  - Chang Gong Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
- The National Children's Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries, aggregate data and analytical plan can be shared with investigators who submit their requests to the Responsible Party with a reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Start Date: December 2028 End Date: December 2029
Access Criteria: Researchers should submit the request to the Responsible Party listed in this study. Data dictionaries, aggregate data and analytical plan can be shared.

REFERENCES:
- [Background] Arabi YM, Alsaawi A, Alzahrani M, Al Khathaami AM, AlHazme RH, Al Mutrafy A, Al Qarni A, Vishwakarma RK, Al Anazi R, Al Qasim E, Abdukahil SA, Al-Rabeah FK, Al Ghamdi H, Alatassi A, Al-Dorzi HM, Al-Hameed F, Babakr R, Alghamdi AA, Bin Salih S, Alharbi A, AlKatheri ME, Mustafa H, Al-Qahtani S, Al Qahtani S, Alselaim N, Tashkandi N, Alyami AH, Alyousef Z, AlDibasi O, Al-Qahtani AH, Aldawood A, Caswell A, Al Ayadhi N, Al Rehaili H, Al Arfaj A, Al Mubarak H, Alwasaidi T, Zahrani S, Alalawi Y, Alhadab A, Nasser T, Omer T, Al Johani SM, Alajlan A, Sadat M, Alzunitan M, Al Mohrij S; SCREEN Trial Group and the Saudi Critical Care Trials Group. Electronic Sepsis Screening Among Patients Admitted to Hospital Wards: A Stepped-Wedge Cluster Randomized Trial. JAMA. 2025 Mar 4;333(9):763-773. doi: 10.1001/jama.2024.25982. PMID 39658862
- [Background] Sanchez-Pinto LN, Bennett TD, DeWitt PE, Russell S, Rebull MN, Martin B, Akech S, Albers DJ, Alpern ER, Balamuth F, Bembea M, Chisti MJ, Evans I, Horvat CM, Jaramillo-Bustamante JC, Kissoon N, Menon K, Scott HF, Weiss SL, Wiens MO, Zimmerman JJ, Argent AC, Sorce LR, Schlapbach LJ, Watson RS; Society of Critical Care Medicine Pediatric Sepsis Definition Task Force; Biban P, Carrol E, Chiotos K, Flauzino De Oliveira C, Hall MW, Inwald D, Ishimine P, Levin M, Lodha R, Nadel S, Nakagawa S, Peters MJ, Randolph AG, Ranjit S, Souza DC, Tissieres P, Wynn JL. Development and Validation of the Phoenix Criteria for Pediatric Sepsis and Septic Shock. JAMA. 2024 Feb 27;331(8):675-686. doi: 10.1001/jama.2024.0196. PMID 38245897
- [Background] Schlapbach LJ, Weiss SL, Bembea MM, Carcillo JA, Leclerc F, Leteurtre S, Tissieres P, Wynn JL, Zimmerman J, Lacroix J; Pediatric Organ Dysfunction Information Update Mandate (PODIUM) Collaborative. Scoring Systems for Organ Dysfunction and Multiple Organ Dysfunction: The PODIUM Consensus Conference. Pediatrics. 2022 Jan 1;149(1 Suppl 1):S23-S31. doi: 10.1542/peds.2021-052888D. PMID 34970683
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Watson RS, Carrol ED, Carter MJ, Kissoon N, Ranjit S, Schlapbach LJ. The burden and contemporary epidemiology of sepsis in children. Lancet Child Adolesc Health. 2024 Sep;8(9):670-681. doi: 10.1016/S2352-4642(24)00140-8. PMID 39142741
- [Background] Schlapbach LJ, Watson RS, Sorce LR, Argent AC, Menon K, Hall MW, Akech S, Albers DJ, Alpern ER, Balamuth F, Bembea M, Biban P, Carrol ED, Chiotos K, Chisti MJ, DeWitt PE, Evans I, Flauzino de Oliveira C, Horvat CM, Inwald D, Ishimine P, Jaramillo-Bustamante JC, Levin M, Lodha R, Martin B, Nadel S, Nakagawa S, Peters MJ, Randolph AG, Ranjit S, Rebull MN, Russell S, Scott HF, de Souza DC, Tissieres P, Weiss SL, Wiens MO, Wynn JL, Kissoon N, Zimmerman JJ, Sanchez-Pinto LN, Bennett TD; Society of Critical Care Medicine Pediatric Sepsis Definition Task Force. International Consensus Criteria for Pediatric Sepsis and Septic Shock. JAMA. 2024 Feb 27;331(8):665-674. doi: 10.1001/jama.2024.0179. PMID 38245889